CLINICAL TRIAL: NCT01245894
Title: Effect of Intensive Lipid Lowering Treatment Compared to Moderate Lipid Lowering Treatment on the Coronary Microcirculation
Brief Title: Influence of Intensive Lipid Lowering Treatment Compared to Moderate Lipid Lowering Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: MD Rasmus Egede, Department of Cardiology, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VF-20060
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2007-11

CONDITIONS: Myocardial Infarction [C14.907.585.500]
Keywords: Index of microcirculatory resistance; Fractional Flow Reserve
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose Rosuvastatin (Active Comparator): 5mg Rosuvastatin/day
  Interventions: Drug: Low-dose Rosuvastatin
- High-dose Rosuvastatin (Active Comparator): Rosuvastatin 40mg/day
  Interventions: Drug: High-dose Rosuvastatin

INTERVENTIONS:
Drug: Low-dose Rosuvastatin — Rosuvastatin 5mg/day for one year
  Other Names: Crestor
  Arms: Low-dose Rosuvastatin
Drug: High-dose Rosuvastatin — Rosuvastatin 40mg/day for one year
  Other Names: Crestor
  Arms: High-dose Rosuvastatin

SUMMARY:
The aim of this study was to measure the effect of low- and high-dose lipid-lowering treatment with rosuvastatin on the coronary physiology parameters.

ELIGIBILITY:
Inclusion Criteria:

1. ST-segment elevation myocardial infarction
2. no prior treatment with statins and
3. a non significant lesion in one of the two non-culprit coronary arteries

Exclusion Criteria:

1. age below 18 or above 81 years,
2. unconscious patients,
3. serum creatinine > 176μmol/L,
4. hypothyroidism ((TSH > 1.5 x ULN (upper limit of normal)),
5. current liver disease (ALAT > 2 x ULN),
6. unexplained creatine kinase > 3 x ULN,
7. alcohol or drug abuse within the last five years,
8. prior myopathy or serious hypersensitivity reaction caused by statins,
9. women with childbearing potential who were not using chemical or mechanical contraception,
10. pregnant or breastfeeding women,
11. history of malignancy unless a disease-free period of more than five years was present,
12. patients with abnormal lung function test (LFT),
13. participation in another investigational drug study less than four weeks before enrolment in the present study,
14. treatment with cyclosporine or fibrates

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the change from baseline in Index of microcirculatory resistance(IMR). | One year

SECONDARY OUTCOMES:
The secondary endpoints were the changes from baseline in Fractional Flow Reserve (FFR) and lipid values. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Egede, MD, Principal Investigator — Department of Cardiology, Odense University Hospital
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Fuenen, Denmark